CLINICAL TRIAL: NCT06886997
Title: Pelvic Floor Ultrasound Versus Urodynamic Studies in Evaluating Women With Stress Urinary Incontinence
Brief Title: PFU vs. UDS in SUI
Acronym: UDS - PFU
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Salma Salah Eltounsi, Trainee, Ain Shams University
Other Study IDs: UDS-PFU
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-03

CONDITIONS: Stress Urinary Incontinence (SUI)
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Urodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Pelvic Floor Ultrasound — Pelvic Floor Ultrasound will be carried out by a sonographer expert in the technique and who will be blinded from the data of clinical examination as well as the UDS results. The 3D/4D abdominal ultrasound probe will be used to perform a transperineal scan to capture midsagittal pelvic floor views. The test will be conducted both at resting state and during the maximum Valsalva maneuver.
Diagnostic Test: Urodynamic studies — Urodynamic studies (UDS) will be carried out according to the usual protocol and will include: cystometry, Valsalva leak point pressure, urethral pressure profile, and uroflowmetry.

SUMMARY:
The goal of this observational stury is to test the diagnostic accuracy of Pelvic Floor Ultrasound in evaluating women with stress urinary incontinence compared to the reference standard Urodynamic Studies. The main question it aims to answer is:

Is Pelvic floor ultrasound as accurate as urodynamic studies in diagnosis of stress urinary incontinence?

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years

Exclusion Criteria:

* Medical history of neurological disorders, cognitive disorders, dementia, Alzheimer's disease, or uncontrolled DM.
* Surgical history of continence or prolapse procedure.
* Examination showing anterior or middle compartment decent with POP-Q staging greater than stage 1, or urogenital fistula.
* Known lower urinary tract or genital tract anomalies or tumors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult women complaining of stress urinary incontinence
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of pelvic floor ultrasound in assessment of stress urinary incontinence compared to urodynamic testing. | Within a week of UDS appointment
  Key Measurements in PFU:
  Bladder neck position at resting and Valsalva states. Bladder Neck Mobility Posterior vesicourethral angle Urethral inclination angle Distance from the external urethral orifice to the bladder neck at resting state.
  Bladder Neck Funneling (BNF)
  Key Parameters Measured in Urodynamics:
  Presence or absence of SUI Presence or absence of Detrusor Overactivity leak point pressure
  Diagnostic accuracy will be assessed according to (sensitivity, specificity, positive and negative predictive values) of PFU compared to UDS (as the gold standard)

SECONDARY OUTCOMES:
Patient satisfaction | Within a week of UDS appointment
  Patient satisfaction by asking which test would she prefer to repeat if needed: the urodynamic study, pelvic floor sonography, or neither?
Cost | Within a week of UDS appointment
  Cost in Egyptian Pounds EGP

REFERENCES:
- [Background] Yao M, Simoes A. Urodynamic Testing and Interpretation. 2023 Aug 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK562310/ PMID 32965981
- [Background] Pietrus M, Pitynski K, Socha MW, Gawron I, Biskupski-Brawura-Samaha R, Waligora M. Enhanced Non-Invasive Diagnosis of Female Urinary Incontinence Using Static and Functional Transperineal Ultrasonography. Diagnostics (Basel). 2024 Nov 14;14(22):2549. doi: 10.3390/diagnostics14222549. PMID 39594215
- [Background] Malmur M, Mlodawski J, Mlodawska M, Misiek M, Adamczyk-Gruszka O, Niziurski P, Gluszek S, Rokita W. Could pelvic floor sonography be a standalone method for excluding genuine stress urinary incontinence in women? Ginekol Pol. 2023 Mar 17. doi: 10.5603/GP.a2023.0026. Online ahead of print. PMID 36929790
- [Background] Lugo T, Leslie SW, Mikes BA, Riggs J. Stress Urinary Incontinence. 2024 Aug 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK539769/ PMID 30969591
- [Background] Hu Y, Lou YL, Zhu SX, Zhang H, Huang T, Wu H, Xie LP. Pelvic floor ultrasound versus urodynamics in evaluating insensible urinary incontinence: A retrospective study. Prog Urol. 2023 Jul;33(7):384-392. doi: 10.1016/j.purol.2023.05.002. Epub 2023 Jun 2. PMID 37271669
- [Background] Dietz HP. Pelvic Floor Ultrasound: A Review. Clin Obstet Gynecol. 2017 Mar;60(1):58-81. doi: 10.1097/GRF.0000000000000264. PMID 28005595
- [Background] Dietz HP. Pelvic floor ultrasound in incontinence: what's in it for the surgeon? Int Urogynecol J. 2011 Sep;22(9):1085-97. doi: 10.1007/s00192-011-1402-7. Epub 2011 Apr 22. PMID 21512829
- [Background] Bahrami S, Khatri G, Sheridan AD, Palmer SL, Lockhart ME, Arif-Tiwari H, Glanc P. Pelvic floor ultrasound: when, why, and how? Abdom Radiol (NY). 2021 Apr;46(4):1395-1413. doi: 10.1007/s00261-019-02216-8. PMID 31529202